CLINICAL TRIAL: NCT02034188
Title: Feasibility Study of Human Umbilical Cord Tissue-Derived Mesenchymal Stem Cells in Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Translational Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBS-UCMSC-001
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; umbilical cord; mesenchymal; stem cells
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Umbilical cord mesenchymal stem cells (Experimental)
  Interventions: Biological: Umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: Umbilical cord mesenchymal stem cells

SUMMARY:
Allogeneic human umbilical cord tissue-derived stem cells injected intravenously (IV) once per day for 7 days is a safe and will induce a therapeutic effect in multiple sclerosis (MS) patients.

DETAILED DESCRIPTION:
The proposed study will assess primarily safety and secondary efficacy endpoints of allogeneic umbilical cord mesenchymal stem cells (UC-MSC) administered to 20 patients with MS.

The primary objective of the trial is freedom from treatment associated adverse events at 4,12 and 52 weeks post treatment. Secondary objective will be efficacy as assessed at baseline, week 12 and 52 and will be quantified based on the following: Neurological assessment of the MS functional composite assessment which comprises of Expanded Disability Status Scale (EDSS), the expanded EDSS (Rating Neurologic Impairment in Multiple Sclerosis, the Scripps neurological rating scale (NRS), paced auditory serial addition test (PASAT), the nine-hole peg test, and 25-foot walking time. Short-form 36 (SF-36) quality of life questionnaire and gadolinium enhanced MRI scans of the brain and cervical spinal cord will also be performed at the indicated time points.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to sign informed consent and capable of understanding the features of this clinical trial.
* Willing to keep a weekly diary and undergo observation for 12 months
* Non-pregnant patients 18-55 years of age with MS according to the revised McDonald criteria and meeting the Poser criteria for clinically defined MS.
* EDSS scores of 2·0 to 5·5 points assessed at least 3 months after the last acute attack of MS.
* Must have proof of health insurance in country of residence.

Exclusion Criteria:

* Patients with evidence of active proliferative retinopathy.
* Patients with poorly controlled diabetes mellitus (glycated hemoglobin: HbA1C > 8.5%).
* Patients with renal insufficiency (Creatinine> 2.5) or failure.
* Infection as evidenced by white blood cell (WBC) count of >15,000 k/cumm and/or temperature > 38 Celsius.
* History of organ transplant.
* History of previous or active malignancy, except for localised cutaneous basal or squamous cell carcinoma or carcinoma in situ of the cervix
* Exercise limiting angina ( Canadian Cardiovascular Society Class 3
* Congestive heart failure (New York Heart Association class 3
* Unstable angina
* Acute ST elevation myocardial infarction (MI) within 1month
* Transient ischemic heart attack or stroke within 1 month
* Severe valvular heart disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 12 months

SECONDARY OUTCOMES:
Number of participants with a change in disability as measured by Expanded Disability Status Scale (EDSS) | 12 months
Number of participants with a change in neurological impairment as measured by Scripps Neurological Rating Scale | 12 months
Number of participants with a change in cognitive function as measured by the • Paced Auditory Serial Addition Test (PASAT) | 12 months
Number of participants with a change in upper extremity function as measured by the Nine Hole Peg Test | 12 months
Number of participants with a change in mobility and leg function as measured by the 25 foot walking test | 12 months
Number of participants with a change in quality of life as measured by the Short form 36 (SF-36) quality of life questionnaire | 12 months
Number of participants experiencing pulmonary edema as measured by 12-lead electrocardiogram (ECG) | 1 month, 3 months
Number of participants with a change in brain or spinal cord lesions as measured by gadolinium-enhanced magnetic resonance imaging (MRI) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Paz-Rodriguez, MD, Principal Investigator — Translational Biosciences / Stem Cell Institute
Locations (1):
- Stem Cell Institute, Panama City, Panama

REFERENCES:
- [Derived] Riordan NH, Morales I, Fernandez G, Allen N, Fearnot NE, Leckrone ME, Markovich DJ, Mansfield D, Avila D, Patel AN, Kesari S, Paz Rodriguez J. Clinical feasibility of umbilical cord tissue-derived mesenchymal stem cells in the treatment of multiple sclerosis. J Transl Med. 2018 Mar 9;16(1):57. doi: 10.1186/s12967-018-1433-7. PMID 29523171